CLINICAL TRIAL: NCT07338383
Title: An Efficacy and Feasibility Trial of a Portable Near Infra-Red Hematoma Imager for Detection of Intracranial Hemorrhage in the Acute Care Setting
Brief Title: Efficacy and Feasibility Trial of a Portable Near Infra-Red Hematoma Imager (NIRD-HI)
Acronym: NIRD-HI
Status: Not yet recruiting | Type: Observational
Sponsor: The Geneva Foundation (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C.2026.013; RC240162 (Other: CDMRP-eBRAP Log Number)
Record Dates: First submitted 2025-12-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury; Intracranial Hemorrhages; Combat Casualty Care; Point of Care
Keywords: Traumatic Brain Injury; Intracranial Hemorrhage; NIRD-HI
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 40 participants with positive head bleed on CT report: Subjects with positive head CT reports that may have a diagnosis of TBI or intracranial hemorrhage
  Interventions: Diagnostic Test: NIRD-HI scan at the time of enrollment; Diagnostic Test: Secondary NIRD-HI scan when a planned repeat CT is performed
- 40 participants with negative head bleed on CT report: Subjects without positive head CT reports that may have a diagnosis of TBI or intracranial hemorrhage
  Interventions: Diagnostic Test: NIRD-HI scan at the time of enrollment; Diagnostic Test: Secondary NIRD-HI scan when a planned repeat CT is performed

INTERVENTIONS:
Diagnostic Test: NIRD-HI scan at the time of enrollment — All enrolled patients who meet the study's eligibility criteria will receive one NIRD-HI scan at the time of enrollment.
Diagnostic Test: Secondary NIRD-HI scan when a planned repeat CT is performed — For patients requiring a planned repeat CT, a secondary NIRD-HI scan may be performed before the subsequent CT imaging.

SUMMARY:
Traumatic Brain Injury (TBI) is a leading cause of death and disability among military personnel, Veterans, and civilians. One of the most dangerous complications of moderate-to-severe TBI is intracranial hemorrhage (ICH). If not identified and treated promptly, ICH can rapidly lead to worsening neurological damage or death. Current diagnostic tools, such as CT scans, are highly effective but impractical for battlefield or resource-limited environments due to their large size and infrastructure dependency.

The Near-Infrared Detection-Head Imaging (NIRD-HI) system is an innovative, noninvasive device using Near-Infrared Spectroscopy (NIRS) to identify abnormal blood accumulation. Unlike traditional tools, NIRD-HI is compact, lightweight, and portable, making it suitable for remote or austere settings. By dynamically imaging the brain, it generates 3D visualizations that pinpoint the size and location of bleeds, including complex bilateral injuries. This offers a significant improvement over current point-of-injury technologies that lack the resolution to reliably diagnose all forms of ICH.

This study supports the FY24 Combat Readiness Medical Research Program by advancing battlefield diagnostic and triage capabilities. The research will:

* Evaluate NIRD-HI's accuracy compared to CT imaging.
* Assess feasibility in real-world acute care settings.
* Investigate its ability to monitor changes in ICH over time.

These objectives address the military's need for tools that improve rapid diagnosis and decision-making during emergencies. Implementing this research can revolutionize TBI management. For Service Members, NIRD-HI promises a field-ready solution for early detection, enabling faster intervention and more effective triage. By reducing diagnostic delays, it could save lives and prevent long-term complications. Furthermore, the system supports prolonged field care by providing continuous monitoring of evolving injuries.

The benefits extend to civilian healthcare, particularly in rural or underserved areas lacking advanced imaging. This accessibility can improve trauma care outcomes for millions, reduce the burden on healthcare systems, and provide equitable distribution of life-saving technology. By addressing gaps in battlefield medicine, this project aims to enhance medical readiness and improve survivability in the most challenging environments.

DETAILED DESCRIPTION:
Traumatic Brain Injury [TBI] has become the hallmark injury of modern warfare and remains one of the most challenging conditions to diagnose in forward-deployed care settings. One of the primary obstacles in diagnosing TBI on the battlefield is the "silent" or delayed onset of neurological symptoms, which can mask the severity of the injury. A key contributor to poor outcomes in moderate to severe TBI is the presence of acute intracranial bleeding, which can swell rapidly, leading to secondary brain damage or death. Early identification of such bleeds is critical for improving patient survival and neurological recovery.

Currently, CT is the gold standard for diagnosing intracranial hemorrhage [ICH], providing the accuracy needed to detect and evaluate brain bleeds. However, the logistical requirements of CT imaging pose significant challenges in deployed or resource-limited environments. These demands render CT impractical for field use, leaving forward-operating medical personnel without a reliable imaging solution for rapid TBI diagnosis. Consequently, there is a pressing need for portable, point-of-injury [POI] diagnostic tools that can effectively detect brain injuries in austere settings.

In both military and civilian contexts, there is an unmet need for a diagnostic device that can alert medical personnel to changes in ICH status without relying on resource-intensive serial imaging or neurological monitoring. Such a tool could enable timely triage and inform critical medical evacuation decisions, improving outcomes for patients with TBI. Existing POI technologies, however, predominantly rely on functional assessments and indirect measures of TBI, which are inherently subjective and often lack specificity. The reliance on such methods can result in false positives or negatives, particularly in low-incidence injuries, where positive predictive value [PPV] tends to fall below 50%. In military medicine, ensuring high sensitivity and specificity is crucial, as initiating unnecessary treatment or evacuations can impose significant operational risks and resource costs. A field-ready diagnostic tool capable of accurately identifying ICH and other TBI complications is therefore essential for improving care in both military and civilian emergency settings.

Existing POI technologies, however, predominantly rely on functional assessments and indirect measures of TBI, which are inherently subjective and often lack specificity. The reliance on such methods can result in false positives or negatives, particularly in low-incidence injuries, where positive predictive value [PPV] tends to fall below 50%. In military medicine, ensuring high sensitivity and specificity is crucial, as initiating unnecessary treatment or evacuations can impose significant operational risks and resource costs. A field-ready diagnostic tool capable of accurately identifying ICH and other TBI complications is therefore essential for improving care in both military and civilian emergency settings.

Near-Infrared Spectroscopy [NIRS] can be used to interrogate tissue. It has been well studied over the years and it can be shown that the principal components of variation in intensity response from tissue can be ascribed to blood volume and oxygenation. The reflected light from the NIR source is used to determine the presence of blood volume in the tissue beneath the sensor. By comparing tissues from different locations within the brain the presence of large volumes of blood that represent a pathological event can be detected. The use of near infra-red [NIR] to estimate the presence of intracranial bleeding spectroscopically has been previously demonstrated, with high agreement with traditional head CT. Though effective for detection of a statichemorrhagic event, there are no currently available NIR-based technology that employs dynamic structural imaging. Moreover, current tools cannot reliably diagnose all types of hematomas, particularly bilateral head injuries.

IMPACT AND RELEVANCE. Approximately 60% of wounded soldiers sustain blast injuries and two-thirds are diagnosed with a TBI. While the majority of TBIs are mild and nonfatal, 17-20% of severe TBI patients die within the first 24 hours after injury underscoring the importance of rapid assessment and accurate triage. Of those who survive the acute phase of a TBI, up to 57% experience chronic health problems related to their injury. This translates to a great economic burden and severe reduction of quality of life for millions of Service Members, Veterans, and civilians. Demonstration of a rapid triage tool for ICH resulting from TBI may expedite diagnosis and treatment, which could minimize the adverse consequences of TBI. Alternatively, the device could rule out injuries for which medical evacuation is non-emergent, preserving Force resources. Advancement of POI diagnostic tools hinges on the demonstration of the efficacy and feasibility of the tool in the acute care setting. In alignment with the goals of conducting high impact translational research that will accelerate innovative ideas into clinical applications that are relevant to Service Members, Veterans, and their families, this study aims to provide critical performance evaluation for the NIRD HI in a US population of TBI patients. Although this study will be conducted in level I trauma center, the questions addressed are applicable to military practice, prolonged field care in particular. Current Joint Trauma System Clinical Practice Guideline [JTS CPG)] for TBI management in prolonged field care [CPG ID: 63] rely on specialized assessments and/or equipment to detect raised intracranial pressure resulting from an ICH. Earlier detection of an intracranial bleed, prior to clinical deterioration, could change triage priorities and inform medical evacuation plans, key to decreasing mortality and improving functional outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 89 years of age
* Able to provide written informed consent either by self or legally authorized representative
* Received head CT imaging on admission
* Able to complete at least one NIRD-HI scan within 4 hours of head CT
* Non-operative management planned

Exclusion Criteria:

* Presence of penetrating or non-survivable injuries
* Hemorrhagic shock or large volume transfusion [>3 units of any blood product within

  1 hour of scan]
* Large open skull wounds, scalp lacerations or surface hematomas prohibiting safe or comfortable sensor placement
* Presence of heat tattoos or intracranial metal fixtures
* Cervical injury prolonging C-spine collar
* Known prisoners or wards of state
* Any condition or finding that makes the patient unsuitable for image acquisition in the Investigator's opinion

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Access to the proposed population includes a mixture of 15% active-duty military and/or VA patients and 85% civilians from central/southern Texas, including the 22 surrounding counties that are receiving trauma care at Brooke Army Medical Center.
  Daily review of the Trauma census will be conducted to review eligible patients. This screening tool will help determine, predict, and address challenges to recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance | Baseline, at time of NIRD-HI testing administered
  Diagnostic Performance. Establish the sensitivity, specificity, PPV, and NPV of the NIRD-HI system for detecting ICH in TBI patients, with a target sensitivity and specificity exceeding 90%.
Feasibility Assessment - Scan Time | Enrollment through study completion, an average of 1 year
  Time in minutes to complete scans in acute care setting recorded on a templated study log including scan start/stop time, interruptions and reasons for interruptions, technical errors and unanticipated device adverse events.
Feasibility Assessment - Operator Usability | Near the end of recruitment period, an average of 1 year
  Operator usability near the end of the recruitment period, 4-6 blinded clinicians (physicians and/or mid-level practritioners) will make a determination of criteria positive or negative research scans assigned in random order to establish statistics for inter-reader agreement. Blinded readers will assign a likelihood score using a Visual Analog Scale [VAS] to indicate how confident they are in their read.
Feasibility Assessment - Device Integration | Enrollment through study completion, an average of 1 year
  Device integration, through operator feedback questionnaire regarding ease of use.
Monitoring of ICH Progression | Baseline, at time of NIRD-HI testing administered
  NIRD-HI readouts for the presence/absence of ICH and region of detection [if positive] as determined by the research device. NIRD-HI readouts will be correlated with Head CT results after each scan.

SECONDARY OUTCOMES:
Diagnostic Performance - Time Detection of ICH | Baseline, at time of NIRD-HI testing administered
  Start/stop times of NIRD-HI readouts will be correlated with Head CT results after each scan for accuracy and start/stop times of scans.
Diagnostic Performance - Operator Performance | Baseline, at time of NIRD-HI testing administered
  Ability to perform NIRD-HI scans [i] scans not performed for subjectreasons [e.g. wounds, bandages, c-spine protection]; [ii] scans not performed for operator reasons [e.g. inability to use device correctly); [iii] scans not performed because of technical issues with the device; and [c] inter-reader agreement.
Accuracy of evolution testing [first NIRD HI scan vs. second NIRD HI] | Baseline, at time of NIRD-HI testing administered
  A subset of subjects with available follow-up head CT will be compared to changes confirmed by CT imaging, to evaluate the efficacy of the device for monitoring intracranial hemorrhages.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Rizzo, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD data will not be shared

REFERENCES:
- [Background] Taylor CA, Bell JM, Breiding MJ, Xu L. Traumatic Brain Injury-Related Emergency Department Visits, Hospitalizations, and Deaths - United States, 2007 and 2013. MMWR Surveill Summ. 2017 Mar 17;66(9):1-16. doi: 10.15585/mmwr.ss6609a1. PMID 28301451
- [Background] Law ZK, Dineen R, England TJ, Cala L, Mistri AK, Appleton JP, Ozturk S, Bereczki D, Ciccone A, Bath PM, Sprigg N; TICH-2 investigators. Predictors and Outcomes of Neurological Deterioration in Intracerebral Hemorrhage: Results from the TICH-2 Randomized Controlled Trial. Transl Stroke Res. 2021 Apr;12(2):275-283. doi: 10.1007/s12975-020-00845-6. Epub 2020 Sep 9. PMID 32902808
- [Background] McCredie VA, Chavarria J, Baker AJ. How do we identify the crashing traumatic brain injury patient - the intensivist's view. Curr Opin Crit Care. 2021 Jun 1;27(3):320-327. doi: 10.1097/MCC.0000000000000825. PMID 33852501
- [Background] Fletcher-Sandersjoo A, Tatter C, Tjerkaski J, Bartek J Jr, Maegele M, Nelson DW, Svensson M, Thelin EP, Bellander BM. Time Course and Clinical Significance of Hematoma Expansion in Moderate-to-Severe Traumatic Brain Injury: An Observational Cohort Study. Neurocrit Care. 2023 Feb;38(1):60-70. doi: 10.1007/s12028-022-01609-w. Epub 2022 Sep 27. PMID 36167951
- [Background] Tien HC, Jung V, Pinto R, Mainprize T, Scales DC, Rizoli SB. Reducing time-to-treatment decreases mortality of trauma patients with acute subdural hematoma. Ann Surg. 2011 Jun;253(6):1178-83. doi: 10.1097/SLA.0b013e318217e339. PMID 21494125
- [Background] Kainerstorfer JM, Ehler M, Amyot F, Hassan M, Demos SG, Chernomordik V, Hitzenberger CK, Gandjbakhche AH, Riley JD. Principal component model of multispectral data for near real-time skin chromophore mapping. J Biomed Opt. 2010 Jul-Aug;15(4):046007. doi: 10.1117/1.3463010. PMID 20799809
- [Background] Robertson CS, Zager EL, Narayan RK, Handly N, Sharma A, Hanley DF, Garza H, Maloney-Wilensky E, Plaum JM, Koenig CH, Johnson A, Morgan T. Clinical evaluation of a portable near-infrared device for detection of traumatic intracranial hematomas. J Neurotrauma. 2010 Sep;27(9):1597-604. doi: 10.1089/neu.2010.1340. PMID 20568959
- [Background] Gramer R, Shlobin NA, Yang Z, Niedzwiecki D, Haglund MM, Fuller AT. Clinical Utility of Near-Infrared Device in Detecting Traumatic Intracranial Hemorrhage: A Pilot Study Toward Application as an Emergent Diagnostic Modality in a Low-Resource Setting. J Neurotrauma. 2023 Aug;40(15-16):1596-1602. doi: 10.1089/neu.2021.0342. Epub 2022 Aug 2. PMID 35856820
- [Background] Riley JD, Amyot F, Pohida T, Pursley R, Ardeshirpour Y, Kainerstorfer JM, Najafizadeh L, Chernomordik V, Smith P, Smirniotopoulos J, Wassermann EM, Gandjbakhche AH. A hematoma detector-a practical application of instrumental motion as signal in near infra-red imaging. Biomed Opt Express. 2012 Jan 1;3(1):192-205. doi: 10.1364/BOE.3.000192. Epub 2011 Dec 20. PMID 22254179
- [Background] Bell RS, Vo AH, Neal CJ, Tigno J, Roberts R, Mossop C, Dunne JR, Armonda RA. Military traumatic brain and spinal column injury: a 5-year study of the impact blast and other military grade weaponry on the central nervous system. J Trauma. 2009 Apr;66(4 Suppl):S104-11. doi: 10.1097/TA.0b013e31819d88c8. PMID 19359953
- [Background] Centers for Disease Control and Prevention, National Center for Injury Prevention and Control. Report to Congress on traumatic brain injury in the United States: Epidemiology and rehabilitation. Atlanta (GA): Centers for Disease Control and Prevention; 2015